CLINICAL TRIAL: NCT04621799
Title: A Prospective Registry Study Evaluating the Safety and Efficacy of Fibrin for Chronic Multi-level Discogenic Low Back Pain
Brief Title: Fibrin for Chronic Multi-level Discogenic Low Back Pain
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pauza, Kevin, MD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Regen_006-0120
Record Dates: First submitted 2020-11-05; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Low Back Pain; Disc Disease; Disc Degeneration; Radiculopathy; Annular Disc Tear
Keywords: Non-autologous fibrin; Minimally Invasive; Injections; Intervertebral disc; Annulus Fibrosus; Sciatica
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration; Radiculopathy; Sciatica | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Intervention Model Description: A prospective evaluation of a cohort of patients with a specific characteristic over time to see if they develop a particular endpoint or outcome based on a stated hypothesis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fibrin Group (Experimental): Experimental: Non-Autologuos Fibrin (NAF) Subjects in the NAF arm received an injection of non-autologous fibrin
  Interventions: Drug: Fibrin sealant

INTERVENTIONS:
Drug: Fibrin sealant — The intra-annular delivery of non-autologous fibrin into the annulus
  Other Names: Baxter Tisseel

SUMMARY:
Intra-annular injections of non-autologous fibrin for moderate to severe chronic low back pain (LBP).

DETAILED DESCRIPTION:
The purpose of this study is to analyze data available in the PIs Regenerative Orthobiologics Registry (ROR) and corresponding patient charts that will either support or refute the efficacy of Intra-annular fibrin as treatment for moderate to severe low back pain. Additionally, we seek to retrospectively identify possible predisposing factors that are correlated with positive outcomes with respect to patient-reported pain and function.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of Intra-annular fibrin injection for annular defects identified radographically and by annulogram

Exclusion Criteria:

* Scoliosis greater than 20 degrees
* Spondylolysis
* Spondylolisthesis greater than Grade 1
* Disc extrusion
* Disc herniations or bulges > 4mm causing severe stenosis
* Prior lumbar surgery or intradiscal procedure (i.e. intradiscal electrothermal therapy, nucleoplasty)
* Cauda equina syndrome
* Active malignancy or tumor as source of symptoms
* Evidence of prior lumbar vertebral body fracture or trauma
* Foraminal stenosis at the affected levels resulting in severe thecal sac compression
* Dynamic instability on lumbar flexion/extension radiographs
* Positive response to diagnostic medial branch block or facet joint injection or sacroiliac joint injection
* Known bleeding disorder
* Known or suspected hypersensitivity or allergy to drugs or components of the fibrin sealant, including aprotinin, used in the procedure
* Presence of ferromagnetic implants that would interfere with MRI evaluations
* Active or pending workers' compensation claims or other litigation related to the condition.
* Pregnant or plans to become pregnant over the course of study participation (2 years)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Two Years
  The Oswestry Disability Index (ODI) is a questionnaire used by clinicians and researchers to quantify disability for low back pain. Scale for the ODI is from 0 (best) - 100 (worst).

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | Two Years
  The NRS consists of a numeric version of the visual analog scale. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible. Scale for NRS is from 0 (best) - 10 (worst).
Visual Analog Scale (VAS) for back pain | Two Years
  When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. Scale for VAS for back pain is from 0 (best) - 10 (worst).
Visual Analog Scale (VAS) for leg pain | Two Years
  When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. Scale for VAS for leg pain is from 0 (best) - 10 (wors
PROMIS Physical Health | Two Years
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. Scale for PROMIS Physical Health is from 16.2 (worst) - 67.7 (best)
PROMIS Mental Health | Two Years
  The PROMIS Global-10 is a publicly available global health assessment tool that allows measurements of symptoms, functioning, and healthcare-related quality of life (HRQoL) for a wide variety of chronic diseases and conditions. Scale for PROMIS Mental Health is from 21.2 (worst) - 67.6 (best).
North American Spine Society (NASS) for patient satisfaction | Two Years
  The North American Spine Society (NASS) developed an outcome assessment instrument to measure diverse dimensions of the impact of lumbar spine problems. Scale range is from 1 to 4 (best to worst).
EURO Quality of Life (EuroQol) | Two Years
  EuroQol is an instrument which evaluates the generic quality of life developed in Europe and widely used. Scale is from 0.33 (worst - 0.88 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Pauza, MD, Principal Investigator — INTERVENTIONAL SPINE SPECIALIST
Locations (1):
- Interventional Spine Specialist, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No